CLINICAL TRIAL: NCT05225233
Title: Transcranial Direct Current Stimulation (tDCS) With Cognitive Training to Reduce Impulsivity and Weight in Veterans With Obesity: A Clinical Trial
Brief Title: tDCS With Cognitive Training to Reduce Impulsivity and Weight in Veterans With Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NURA-009-21S
Record Dates: First submitted 2022-01-19; First posted 2022-02-04 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Obesity
Keywords: transcranial direct current stimulation; neuromodulation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tDCS with Cognitive Training (Experimental): Participants will receive active tDCS stimulation with their cognitive training during a one-hour session each day which includes 20 minutes of stimulation at the beginning of a 46-minute task training session. Ten sessions will be completed over three weeks.
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS with Cognitive Training (Sham Comparator): Participants will receive 10 sessions of cognitive training concurrent with sham tDCS. For sham tDCS, electrodes are placed at the same locations as for active tDCS, but current is ramped up for the initial 30 seconds, then immediately ramped back down. This method mimics the initial physical sensation of stimulation, but there is no active current for the remainder of the session.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Cognitive training concurrent with sham tDCS (30 seconds ramp up/ramp down at the beginning of the session)
  Arms: Sham tDCS with Cognitive Training
Device: Active Transcranial Direct Current Stimulation (tDCS) — Cognitive training concurrent with 2 mAmps of anodal stimulation applied to the left frontal cortex for 20 minutes.
  Arms: Active tDCS with Cognitive Training

SUMMARY:
The purpose of this study is to investigate if transcranial direct current stimulation (tDCS) can increase the effectiveness of cognitive training to reduce impulsivity in individuals with obesity, and to evaluate weight change with these individuals. The long-term goal of this research is to develop new treatment approaches for individuals with obesity.

DETAILED DESCRIPTION:
Two-hundred forty individuals will be screened with the goal of consenting and enrolling up to 124 patients and 88 patients completing the study. Participants completing the study will concurrently complete a structured weight loss program. The investigators' study protocol will consist of 13 study visits including four testing days, one before (V1), one on the day of the tenth session of tDCS (V11), another test visit (V12) 6 weeks later, and a final test visit approximately 4 months after beginning stimulation (V13).

ELIGIBILITY:
Inclusion Criteria:

* Veteran enrolled in a MOVE! Weight Management Program (group or individual) at the Minneapolis VA Health Care System
* Obese (BMI>30 or BMI>27 plus at least one weight-related comorbidity)
* Adults, ages 18 years or older (up to age 80)
* Able to understand English, self-consent and follow study-related procedures
* Willing to use a reliable form of birth control if they are of females of child-bearing potential

Exclusion Criteria:

* History of any of the following: seizures, severe or moderate head injury, head surgery, significant neurological disorder (significance based on Principal Investigator's judgment)
* Frequent severe headaches
* History of scalp conditions such as eczema or seborrheic dermatitis
* Metal in head (other than in mouth) including shrapnel/surgical clips/welding fragments
* Implanted medical devices (including pumps and cardiac pacemakers)
* Pregnancy
* Acute substance dependence or withdrawal that would affect ability to complete cognitive training
* Moderately severe to severe depression (as identified on PHQ-9 scale during baseline screening)
* Other psychological or medical disorders requiring inpatient treatment (as identified during chart review)
* Presence of a known metabolic or hormonal disorder (such as Cushing's, untreated thyroid dysfunction, or uncontrolled diabetes mellitus defined as a hemoglobin A1c > 8.0), or significant edema/volume overload - all of which would affect weight
* Uncontrolled hypothyroidism that would affect weight

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in task impulsivity as measured by the NIH Flanker | Change between baseline and Visit 11, Visit 12 (approximately 2 months), and Visit 13 (approximately 4 months)
  Differences in the magnitude of change in NIH Flanker Reaction Time (RT) (ms) between active and sham groups from baseline to follow up sessions.
Change in weight | Change between baseline and Visit 12 (approximately 2 months), and Visit 13 (approximately 4 months)
  Differences in the magnitude of change in weights (kg) between active and sham tDCS (active from baseline to follow up sessions.

SECONDARY OUTCOMES:
Change in reported impulsivity as measured by the Barratt Impulsiveness Scale (BIS) | Change between baseline and Visit 11, Visit 12 (approximately 2 months), and Visit 13 (approximately 4 months)
  Differences in the magnitude of change in BIS scores (Likert scale points) will be compared between active and sham tDCS groups from baseline to follow up sessions.
Change in reported impulsivity as measured by the UPPS-P Impulsive Behavior Scale (UPPS-P) | Change between baseline and Visit 11, Visit 12 (approximately 2 months), and Visit 13 (approximately 4 months)
  Differences in the magnitude of change in UPPS-P scores (Likert scale points) will be compared between active and sham tDCS groups from baseline to follow up sessions.
Change in reported binge eating as measured by the Binge Eating Scale (BES) | Change between baseline and Visit 11, Visit 12 (approximately 2 months), and Visit 13 (approximately 4 months)
  Differences in the magnitude of change in BES scores (Likert scale points) will be compared between active and sham tDCS groups from baseline to follow up sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Shalamar D Sibley, MD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No